CLINICAL TRIAL: NCT03875183
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of INL1 in Patients With Heart Failure and Reduced Ejection Fraction
Brief Title: Study to Evaluate Effects of INL1 in Patients With Heart Failure and Reduced Ejection Fraction
Acronym: TRACER-HF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innolife Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INL1-001; 2019-000511-89 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Reduced Ejection Fraction
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INL1 50mg BID (Experimental): INL1 50mg dose to be given twice daily using one 50mg capsule and two matching placebo capsules at each dose
  Interventions: Drug: INL1
- INL1 150 mg BID (Experimental): INL1 150mg dose to be given twice daily using three 50mg capsules at each dose
  Interventions: Drug: INL1
- INL1 300 mg BID (Experimental): INL1 300mg dose to be given twice daily using three 100mg capsules at each dose
  Interventions: Drug: INL1
- Placebo (Placebo Comparator): Placebo dose to be given twice daily using 3 placebo capsules at each dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INL1 — Capsules
  Arms: INL1 150 mg BID; INL1 300 mg BID; INL1 50mg BID
Other: Placebo — Capsules
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-response trial in patients with chronic stable Heart Failure (HF) and reduced Left Ventricular Ejection Fraction (LVEF) to evaluate the efficacy and safety of three INL1 doses compared with placebo. Patients will be treated for approximately 12 weeks with one of three INL1 doses: 50 mg, 150 mg, 300 mg, or, placebo capsules, taken twice daily (BID).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HF requiring chronic treatment of loop diuretics
* Left Ventricular Ejection Fraction (LVEF) ≤ 40% at screening by echocardiography
* N-Terminal-prohormone of Brain Natriuretic Peptide (NT-proBNP) ≥400 pg/mL at screening for patients without atrial fibrillation or atrial flutter, or, NT-proBNP ≥ 1,200 pg/mL at screening for patients with atrial fibrillation or atrial flutter
* Treated for Heart Failure with stable, optimal pharmacological therapy
* Acceptable screening echocardiographic image quality

Exclusion Criteria:

* Female patients of childbearing potential
* Patients with a New York Heart Association (NYHA) Class I or IV
* Heart failure that is clearly caused by toxin / drug such as Adriamycin
* Significant medical conditions or recent history suggesting the patient's study participation will potentially pose a major risk to patient's safety and well-being
* Need for routine scheduled outpatient IV infusions for Heart Failure or scheduled ultrafiltration
* History of rhabdomyolysis or history of autoimmune diseases
* Severe renal disease
* Hepatic disease
* Pulmonary disease limiting exercise capacity
* Atrial fibrillation with rapid ventricular response
* Life expectancy of less than 6 months
* Type 1 diabetes mellitus or Type 2 diabetes mellitus with very poor glycemic control
* Patients with anemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Proportional change in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | Baseline - 12 weeks
  Proportional change in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) from Baseline to 12 weeks

SECONDARY OUTCOMES:
Composite Heart Failure (HF) Improvement Score | Baseline - 12 weeks
  Composite HF Improvement Score, summarizing changes in 4 HF outcomes (NT-proBNP, left ventricular end-systolic volume [LVESV], NYHA class, and 6 Minute Walk Test) from Baseline to 12 weeks
Change in Left Ventricular End Diastolic (LVED) | Baseline - 12 weeks
  Echocardiogram finding: change in LVED from Baseline to 12 weeks
Change in Left Ventricular End Systolic (LVES) | Baseline - 12 weeks
  Echocardiogram finding: change in LVES from Baseline to 12 weeks
Change in Left Ventricular End Diastolic Volume (LVEDV) | Baseline - 12 weeks
  Echocardiogram finding: change in LVEDV from Baseline to 12 weeks
Change in Left Ventricular End Systolic Volume (LVESV) | Baseline - 12 weeks
  Echocardiogram finding: change in LVESV from Baseline to 12 weeks
Change in Left Ventricular Systolic Volume (LVSV) | Baseline - 12 weeks
  Echocardiogram finding: change in LVSV from Baseline to 12 weeks
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline - 12 weeks
  Echocardiogram finding: change in LVEF from Baseline to 12 weeks
Change in Left Ventricular Mass (LVM) | Baseline - 12 weeks
  Echocardiogram finding: change in LVM from Baseline to 12 weeks
Change in Left Ventricular End Diastolic Diameter (LVEDD) | Baseline - 12 weeks
  Echocardiogram finding: change in LVEDD from Baseline to 12 weeks
Change in Left Ventricular End Systolic Diameter (LVESD) | Baseline - 12 weeks
  Echocardiogram finding: change in LVESD from Baseline to 12 weeks
Change in Left Ventricular Fractional Shortening (LVFS) | Baseline - 12 weeks
  Echocardiogram finding: change in LVFS from Baseline to 12 weeks
Change in ratio of mitral peak velocity of early filling (E) to early diastolic mitral annular velocity (E') | Baseline - 12 weeks
  Echocardiogram finding: change in E/E' ratio from Baseline to 12 weeks
Change in Left Atrial Volume (LAV) | Baseline - 12 weeks
  Echocardiogram finding: change in LAV from Baseline to 12 weeks
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) | Baseline - 12 weeks
  Echocardiogram finding: change in TAPSE from Baseline to 12 weeks
Change in Tricuspid Regurgitation (TR) peak velocity | Baseline - 12 weeks
  Echocardiogram finding: change in TR peak velocity from Baseline to 12 weeks
Change in Tricuspid Regurgitation (TR) gradient | Baseline - 12 weeks
  Echocardiogram finding: change in TR gradient from Baseline to 12 weeks
Change in Tricuspid Regurgitation (TR) severity | Baseline - 12 weeks
  Echocardiogram finding: change in TR severity from Baseline to 12 weeks
Change in Inferior Vena Cava (IVC) Diameter | Baseline - 12 weeks
  Echocardiogram finding: change IVC Diameter from Baseline to 12 weeks
Change in New York Heart Association (NYHA) class | Baseline to 12 weeks
  Change in NYHA class from Baseline to 12 weeks
Change in 6 minute walk distance | Baseline to 12 weeks
  Change in 6 minute walk distance from Baseline to 12 weeks
Quality of Life (QoL) based on Kansas City Cardiomyopathy Questionnaire (KCCQ) change | Baseline to 12 weeks
  QoL based on change in KCCQ from Baseline to 12 weeks. Quality of Life scale can range from 0 to 100, with higher values indicating a better outcome. Change will be calculated by subtraction.
Time to earliest event among the composite of cardiovascular (CV) death, hospitalization for HF, and unplanned use of intravenous diuretics or intensification of oral diuretic dose | Baseline to 12 weeks
  Time to earliest event among the composite of CV death, hospitalization for HF, and unplanned use of intravenous diuretics or intensification of oral diuretic dose from Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chen, MD, Study Chair — Innolife Co., Ltd.
Locations (13):
- United States (12):
  - UCLA School of Medicine, Torrance, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Grady Clinical Research Center, Atlanta, Georgia
  - Via Christi Research, a division of Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Clinical Trials of America LA, LLC, Monroe, Louisiana
  - St Louis Heart and Vascular, St Louis, Missouri
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - East Texas Cardiology, Houston, Texas
  - Angiocardiac Care of Texas, Houston, Texas
- Chongqing University 3 Gorges Hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No